CLINICAL TRIAL: NCT04334044
Title: Treatment of Severe Acute Respiratory Syndrome Caused by COVID-19 With Ruxolitinib
Brief Title: Treatment of SARS Caused by COVID-19 With Ruxolitinib
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grupo Cooperativo de Hemopatías Malignas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAL 345/2020
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: COVID-19; Severe Acute Respiratory Syndrome Coronavirus 2
MeSH Terms: conditions — COVID-19 | interventions — ruxolitinib

STUDY DESIGN:
Intervention Model Description: Use of ruxolitinib on patients with respiratory distress and pneumonia changes on chest computed tomography
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib (Experimental): Ruxolitinib 5 mg BID since the beginning of dyspnea or increment of work of breathing with pneumonia changes in chest CT-scan
  Interventions: Drug: Ruxolitinib Oral Tablet

INTERVENTIONS:
Drug: Ruxolitinib Oral Tablet — Ruxolitinib 5 mg twice a day

SUMMARY:
In December 2019, a new virus emerged in Wuhan, China rapidly becoming a pandemic with registered cases above 800,000 around the world. The virus is now known as SARS-CoV2 calling its disease coronavirus-19 or COVID-19. The mortality of the virus has been reported around 2-10% and its causes because of the proinflammatory immune response generated on the host. The cytokines involved in the immune response to COVID-19 are IL-1, IL-2, IL4, IL-6, IL-10, IL-12, IL-13, IL-17, GCSF, MCSF, IP-10, MCP-1, MIP-1α, HGF, IFN-γ y TNF-α.

Ruxolitinib is an inhibitor of JAK 1/2 which is responsable for multiple cellular signals including the proinflammatory IL-6. Ruxolitinib works as and immunomodulator decreasing the cytotoxic T lymphocytes and increasing the Treg cells.

This study is intended to stop the disregulated immune response caused by COVID-19 that generates the pneumonia and subsequent severe acute respiratory syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed COVID-19 with confirmatory test
* Increase in work of breathing or presence of dyspnea
* Presence of lung changes associated with COVID pneumonia by chest imaging
* Informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding
* Thrombocytopenia below 20,000 cells/mm3
* Neutropenia below 500 cels/mm3
* Known and active infection of HIV, Hepatitis C, Hepatitis B, Herpes Zoster or Mycobacterium Tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Recovery of Pneumonia | 14 days
  Presence of recovery of pneumonia characterized by cease of respiratory symptoms

SECONDARY OUTCOMES:
Response of C-reactive protein | 14 days
  Increment or decrease in mg/ml of C-reactive protein
Response of Ferritin | 14 days
  Increment or decrease in ng/ml of ferritin
Response of D-dimer | 14 days
  Increment or decrease in mg/ml of D-dimer
Rate of ICU admission | 14 days
  Requirement of Intensive Care Unit on the patients under treatment
Rate of mechanical ventilation | 14 days
  Requirement of mechanical ventilation on the patients under treatment
Overall Survival | 1 month
  Time since the diagnosis to the last follow up (recovery or death)
Toxicity Rate | 1 month
  Rate of adverse events associated with ruxolitinib

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo Cooperativo de Hemopatías Malignas, Huixquilucan, State of Mexico, Mexico

IPD SHARING:
Plan to Share IPD: No